CLINICAL TRIAL: NCT05579041
Title: Evaluation of Swallowing Kinematics and Suprahyoid Muscle Activation During Masako, Mendelsohn Maneuvers and Mouth Open Swallowing Maneuver
Brief Title: Compare Swallowing Kinematics and Suprahyoid Muscle Activation Among Three Different Swallowing Tasks
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ömer Faruk Yaşaroğlu, MSc, PT, Hacettepe University
Other Study IDs: MOS Maneuver Kinematic
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to swallowing kinematics and suprahyoid muscle activation among Masako, Mendelsohn Maneuvers and new-designed Mouth Open Swallowing Maneuver

DETAILED DESCRIPTION:
Swallowing disorder can result in aspiration pneumonia, dehydration, malnutrition and even death. Therefore, it is a condition that needs to be detected, prevented and/or treated at an early stage. In the rehabilitation process of swallowing disorders, many exercise approaches are used, as well as compensatory postures and maneuvers. In addition to creating compensation and increasing swallowing muscle strength, the maneuvers used also change the temporal parameters associated with swallowing, such as delay in the swallowing reflex and time to close the airway.

Mendelson maneuver and Masako maneuver are the most commonly used swallowing maneuvers in swallowing rehabilitation. During the Mendelson maneuver, the patient is asked to voluntarily hold larynx when larynx is elevated. Masako maneuver is swallowing with tongue positioned between anterior teeth. Mouth Open Swallowing Maneuver is new-designed exercise. 10 mm wedge is comfortably positioned on the molar teeth and patient is asked to swallow in this way. We think that the explosive force that occurs more hyolaryngeal displacement than normal swallowing. Therefore, The targets of all three exercises in the swallowing physiology is different. It is important to investigate the effects of all three exercises on swallowing physiology in order to determine a patient-specific rehabilitation program and develop new techniques.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Getting less than 3 points from the T-EAT-10 (Turkish Eating Evaluation Questionnaire) questionnaire

Exclusion Criteria:

* Having disc herniation, mechanical neck pain or any pathology in the cervical region.
* Having a temporamandibular joint problem that may affect joint biomechanics and muscle functions.
* Having any neurological or systemic disease,
* Having undergone head and neck surgery or received radiotherapy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult individuals will be included
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Kinematic Analysis | 25 min
  Participants will be asked to perform three repetitions of dry swallowing (control task), Masako and Mendelsohn maneuvers, and Open mouth swallowing exercise during videofluoroscopic swallow study (30 fps) while recording suprahyoid muscle activation simultaneously.

SECONDARY OUTCOMES:
T-EAT 10 questionnaire | 10 min
  T-EAT 10 questionnaire will be made to assess whether participants have swallowing complaints.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demir N, Serel Arslan S, Inal O, Karaduman AA. Reliability and Validity of the Turkish Eating Assessment Tool (T-EAT-10). Dysphagia. 2016 Oct;31(5):644-9. doi: 10.1007/s00455-016-9723-9. Epub 2016 Jul 12. PMID 27405421
- [Result] Azola AM, Greene LR, Taylor-Kamara I, Macrae P, Anderson C, Humbert IA. The Relationship Between Submental Surface Electromyography and Hyo-Laryngeal Kinematic Measures of Mendelsohn Maneuver Duration. J Speech Lang Hear Res. 2015 Dec;58(6):1627-36. doi: 10.1044/2015_JSLHR-S-14-0203. PMID 26426312
- [Result] Byeon H. Effect of the Masako maneuver and neuromuscular electrical stimulation on the improvement of swallowing function in patients with dysphagia caused by stroke. J Phys Ther Sci. 2016 Jul;28(7):2069-71. doi: 10.1589/jpts.28.2069. Epub 2016 Jul 29. PMID 27512266
- [Result] Martin-Harris B, Jones B. The videofluorographic swallowing study. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):769-85, viii. doi: 10.1016/j.pmr.2008.06.004. PMID 18940640
- [Derived] Yasaroglu OF, Serel Arslan S, Cengiz E, Alici R, Demir N, Oguz B, Duger T. Swallowing kinematics and submental muscles activation during a newly designed maneuver called Mouth Open Swallowing Maneuver: A comparative study. PLoS One. 2024 Mar 25;19(3):e0299845. doi: 10.1371/journal.pone.0299845. eCollection 2024. PMID 38527058